CLINICAL TRIAL: NCT07065565
Title: Non-intubated vs Intubated Anesthesia for Tracheal and Carinal Reconstruction
Brief Title: Tubeless Tracheal and Carinal Reconstruction
Acronym: NOVA-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shuben Li (Other)
Responsible Party: Sponsor-Investigator, Shuben Li, Deputy Director, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-2025-075-01
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Tracheal Disease; Airway Disease
Keywords: non-intubated anesthesia; airway disease; tracheal reconstruction; carinal reconstruction
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-intubated group (Experimental): Surgical procedure: non-intubated tracheal and carinal reconstruction
  Interventions: Procedure: non-intubated tracheal and carinal reconstruction
- Intubated group (Active Comparator): Surgical procedure: intubated tracheal and carinal reconstruction
  Interventions: Procedure: intubated tracheal and carinal reconstruction

INTERVENTIONS:
Procedure: non-intubated tracheal and carinal reconstruction — non-intubated tracheal and carinal reconstruction
  Arms: Non-intubated group
Procedure: intubated tracheal and carinal reconstruction — intubated tracheal and carinal reconstruction
  Arms: Intubated group

SUMMARY:
In recent year, non-intubated anesthesia had emerged as an available alternative for thoracic procedure. Whether non-intubated tracheal/carinal reconstruction confers distinct perioperative advantages over the conventional intubated approach remains uncertain. The purpose of this study was to evaluate the safety and perioperative outcomes of non-intubated versus intubated approaches in tracheal and carinal reconstruction.

DETAILED DESCRIPTION:
Tracheal/carinal resection and reconstruction remains a technically demanding procedure with high risks of morbidity and mortality. Traditionally, tracheal surgery is performed under intubated anesthesia, with intermittent endotracheal ventilation to maintain oxygenation during airway reconstruction. However, endotracheal intubation with cross-field ventilation obstructs the surgical field and potentially complicating the reconstruction procedure. Non-intubated anesthesia have has gained widespread adoption for modern thoracic surgery. However, the safety and feasibility of non-intubated tracheal and carinal reconstruction have not been studied by randomized controlled trial. So, this randomized controlled trial aims to evaluate whether the non-intubated approach offers comparable short-term and long-term outcomes to the conventional intubated procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Airway diseases were diagnosed by chest enhanced CT and bronchoscopy
2. The patients with age ≥ 18 and ≤ 80 years old
3. ASA (American Society of Anesthesiologists) stage: I-III
4. sign the informed consent. -

Exclusion Criteria:

1. The patients have proved history of congestive heart failure, angina without good control with medicine; ECG-proved penetrating myocardial infarction; hypertension with bad control; valvulopathy with clinical significance; arrhythmia with high risk and out of control
2. The patients have severe systematic intercurrent disease, such as active infection or poorly controlled diabetes; coagulation disorders; hemorrhagic tendency or under treatment of thrombolysis or anticoagulant therapy
3. Airway anatomical abnormalities due to a history of surgery
4. Patients present with other malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | postoperative in-hospital stay up to 30 days
  The rate of conversion to intubated approach in the operation
Postoperative complications rate | postoperative in-hospital stay up to 30 days
  Number and severity of adverse events that are related to the treatment of each patient. Postoperative treatment-related complications were assessed by the Clavien-Dindo Classification. Treatment-related adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Operative time | postoperative in-hospital stay up to 30 days
  Operative time was defined as the time between the start of the surgery (incision) and the finish of surgery (closure of the skin).
Length of stay (LOS) | postoperative in-hospital stay up to 30 days
  Length of stay is the duration for enrolled patients until the date of meeting the criteria of hospital discharge since the date of surgery.
Postoperative ICU stay | postoperative in-hospital stay up to 30 days
  Postoperative hospital stay is the duration for each patients until the date of meeting the criteria of ICU discharge since the date of surgery.
Intraoperative bleeding loss | postoperative in-hospital stay up to 30 days
  blood loss in the operation
Length of resection | postoperative in-hospital stay up to 30 days
  Length of resection in the operation
Reconstruction time | postoperative in-hospital stay up to 30 days
  Reconstruction time was defined as the time between the start of resection (tracheal) and the finish of reconstruction (tracheal).
Volume of postoperative drainage | postoperative in-hospital stay up to 30 days
  The volume of postoperative drainage of the patient was the sum of his daily drainage volume after the surgery.
1-year disease-free survival (DFS) | 1 year after surgery
  DFS at 1 year after surgery
1-year overall survival(OS) | 1 year after surgery
  OS after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Guangzhou Medical University, Guangdong, Gaungzhou, China

IPD SHARING:
Plan to Share IPD: No